CLINICAL TRIAL: NCT05939024
Title: Efficacy of Conventional Physical Therapy With and Without Muscle Energy Techniques in the Treatment of Chronic Non-Specific Low Back Pain
Brief Title: Efficacy of Muscle Energy Techniques in the Treatment of Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rashid
Record Dates: First submitted 2023-06-20; First posted 2023-07-11 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Low Back Pain, Mechanical
Keywords: Muscle Energy Technique; Physical Therapy; Pain; Functional Disability; Fear Avoidance Beliefs; Quality of Life; Range of Motion
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware of the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy (CPT) Group (Active Comparator): Patients in this group will receive Conventional Physical therapy only, which includes hot pack, TENS, Ultrasonic, stretching and strengthening exercises.
  Interventions: Other: Conventional Physical Therapy
- Muscle Energy Technique plus Conventional Physical Therapy Group (Experimental): In this group, Post Isometric Relaxation of the Muscle Energy Techniques will be applied to the Spinal Stabilizers and Mechanoreceptors in addition to Conventional Physical Therapy.
  Interventions: Other: Muscle Energy Technique plus Conventional Physical Therapy

INTERVENTIONS:
Other: Muscle Energy Technique plus Conventional Physical Therapy — Post-Isometric Relaxation of the Muscle Energy Techniques will be applied to Spinal Stabilizers and Mechanoreceptors. Hold time will be 7 seconds with 5 seconds rest between two performance x 3 times /session. Whereas, Conventional Physical Therapy consists of hot pack, TENS, Ultrasonic along with stretching and exercises of back musculature.
  Other Names: Post-Isometric Relaxation Technique plus Conventional Physical Therapy
  Arms: Muscle Energy Technique plus Conventional Physical Therapy Group
Other: Conventional Physical Therapy — Conventional Physical Therapy consists of hot pack, TENS, Ultrasonic along with stretching and exercises of back musculature.
  Arms: Conventional Physical Therapy (CPT) Group

SUMMARY:
Chronic Non-Specific Low Back Pain is characterized as a tension, soreness and stiffness. Various studies, defined MET as a manual medicine treatment procedure that involves the voluntary contraction of the subject's muscle in a precisely controlled direction, at varying levels of intensity, against a distinctly executed counterforce applied by the therapist.

DETAILED DESCRIPTION:
Chronic Non-specific LBP is located in region below lower costal margins and above inferior gluteal margins with or without any referred pain in legs, an essentially non-attributable to any specific cause. It may lasting for more than 7-12 months and affect individual over a long period of time once in a lifetime at least. METs is useful in increasing extensibility and range of motion of various joints and provides good results in the patients with back pain. These techniques are used as the treatment of weakened muscles, restricted joints, reducing pain reliving muscle tension & spasm, & increased strength of the muscle. MET is a verstile, safe, gentle technique traditionally used to address muscular strain, PAIN, local edema and joint dysfunction. It was reported that post isometric relaxation is considered a highly effective therapy for back dysfunction patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 45 years
2. Gender : both genders
3. Low Back Pain of more than 3 months duration
4. ODI Score between 20-80%
5. BMI: 25-29 Kg/m2
6. VAS: Initial Pain Score > 3
7. Pain Localized to Lower Lumbar Region
8. Decreased Lumbar ROM

Exclusion Criteria:

1. Red Flag Signs of Low Back Pain (Metabolic Bone Disease, Malignancy, Cardiovascular Disorder, Pregnancy)
2. Patient with Paraesthesia or Numbness
3. Disturbed Reflexes (Hypo/Hyper Reflexia)
4. Motor Weakness
5. H/O Low Back Surgery
6. H/O Recent Trauma < 2 Months
7. H/O Rheumatoid Arthritis, Osteoporosis and Fracture
8. Joint hyper mobility.
9. Psychological Mental Disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be measured at the baseline at the time of recruitment, and change in pain intensity will be measured at 2nd week and 3rd week of intervention.
  Pain intensity will be measured using Visual Analogue Scale. It consists of a 10cm line, with two end points, 0 representing no pain and 10 representing pain as bad as it could be possible.
Lumbar Ranges of Motion | Lumbar Range of Motion will be measured at baseline at the time of recruitment and change in range of motion will be measured at 2nd week and 3rd week of treatment.
  Lumbar Ranges of Motion will be measured using inclinometer. The normal amount of lumbar flexion range of motion is 60 degrees, and the normal range of motion of lumbar extension is 25 degrees. The lumbar spine also normally moves 25 degrees in lateral flexion, or side bending.
Functional Disability Level | Level of Functional Disability will be recorded as baseline at the time of recruitment and change in functional status will be observed at the 2nd week and 3rd week of intervention.
  Oswestry Disability Index was used to determine the functional status of individual. The final score ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Change in Fear Avoidance Belief | Fear Avoidance Beliefs will be observed as baseline at the time of recruitment and any change in Fear Avoidance Beliefs will be observed at the 2nd week and 3rd week of treatment.
  Fear Avoidance Beliefs will be observed using Fear Avoidance Beliefs Questionnaire. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Change in Quality of Life | Change in quality of life will be measured at baseline at the time of recruitment and change in quality of life will be measured at the 2nd week and 3rd week of intervention.
  Short Form-36 Health Survey Questionnaire was used to measure change in Quality of Life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Total score of this questionnaire is 100, with lower the score the more disability, the higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr Ashfaq Ahmed, PhD, Study Chair — University of Lahore; Rashid Hafeez Nasir, M. Phil, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Participants data that underlies the results after de-identification
Supporting Information: Study Protocol
Time Frame: Immediately after publication
Access Criteria: Researchers who provide methodological sound proposal